CLINICAL TRIAL: NCT02579928
Title: Efficacy of Rapid-Acting NMDA Antagonist for Treatment of Adolescent Depression and Anxiety Disorders
Brief Title: Ketamine Infusion for Adolescent Depression and Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1506016041
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder; Anxiety Disorder
Keywords: Ketamine; Depression; Major Depressive Disorder; Anxiety; School refusal; Suicide; Generalized Anxiety; Suicidal Ideation
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Depression; Phobia, School; Suicide; Generalized Anxiety Disorder; Suicidal Ideation | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned the treatment order, with participants receiving a single infusion of either ketamine hydrochloride (0.5 mg/kg) or midazolam (0.045 mg/kg) on Day 1, and the alternate compound 2 weeks later.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Midazolam was chosen as an active placebo in keeping with its similar pharmacokinetic profile and precedent as a reasonable comparator for nonspecific behavioral effects of ketamine
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Participants were randomly be assigned to receive a dose of 0.5 mg/kg of Ketamine (administered intravenously over 40 minutes with a maximum total dose allowed in this study will be 50mg).
  Interventions: Drug: Ketamine
- Midazolam (Experimental): Participants were randomly assigned to receive a dose of 0.045mg/kg of Midazolam (administered Intravenously over 40 minutes with a the maximum total dose allowed in this study of 4.5mg),
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — A single dose of 0.5mg/kg of Ketamine will be administered Intravenously during 40 minutes in the Hospital Research Unit of YNHH. The subject will be monitored continuously during the procedure, and every hour for three hours after the infusion.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Midazolam — A single dose of 0.045mg/kg of Midazolam will be administered intravenously during 40 minutes in the Hospital Research Unit of YNHH. The subject will be monitored continuously during the procedure, and every hour for three hours after the infusion.
  Other Names: Versed
  Arms: Midazolam

SUMMARY:
The purpose of this study is to determine the tolerability and short-term efficacy of a single ketamine infusion for the treatment of adolescents with 1) medication-refractory major depressive disorder (MDD) and/or 2) medication-refractory anxiety disorders (social anxiety disorder, panic disorder, generalized anxiety disorder and/or separation anxiety disorder).

DETAILED DESCRIPTION:
We will conduct a crossover trial in which as many as 36 adolescents (18 with MDD and 18 with anxiety disorders) will be given a single infusion of ketamine (study drug) or midazolam (active control). MDD symptoms and anxiety symptoms will be monitored over a two-week period. If applicable, comorbid school refusal symptoms will also be monitored over a two-week period for both cohorts. A 2-week washout period will be required between infusion doses. Our primary outcomes will be 1) improvement in MDD symptoms (measured by Montgomery-Asberg Depression Rating Scale, revised (MADRS) score) 1 day after infusion, for the cohort of subjects enrolled in the MDD arm of this trial and 2) improvement in the anxiety symptoms (measured by the Multimodal Anxiety Scale for Children (MASC) acute physical symptoms subscale) for the cohort of subjects enrolled in the anxiety disorders arm of the trial.

ELIGIBILITY:
Inclusion:

MDD Cohort:

* Meet DSM-5 criteria for Major Depressive Disorder by structured interview (MINI-KID)
* CDRS-R score >40.
* Failure to achieve remission with at least 1 adequate prior antidepressant trial (e.g. SSRI, SNRI, or TCA), meaning at least 8 weeks at therapeutic dosing, including at least 4 weeks of stable dosing.

Anxiety Cohort:

* Meet DSM-5 criteria for any of the following anxiety disorders: Social Anxiety Disorders, Generalized Anxiety Disorder, Separation Anxiety Disorder and/or Panic Disorder by structured interview (MINI-KID)
* ADIS Clinical Severity Rating ≥4 (moderately severe) for any of the 4 included anxiety disorders
* Failure to achieve remission with at least 1 adequate prior anxiolytic medication trial (e.g. SSRI, SNRI, or TCA), meaning at least 8 weeks at therapeutic dosing, including at least 4 weeks of stable dosing.
* Failure to achieve remission with previous CBT or subject declines current CBT therapy

Both cohorts:

* Stable psychiatric medications and doses for the month prior to enrollment. Subjects may continue to engage in any ongoing psychotherapy.
* Medically and neurologically healthy on the basis of physical examination and medical history.
* Parents able to provide written informed consent and adolescents must additionally provide assent.

Exclusion:

* Current inpatient hospitalization or active suicidal ideation requiring referral for inpatient hospitalization for safety.
* History of psychotic disorder or manic episode diagnosed by MINI-KID
* History of substance dependence diagnosis by MINI-KID (excluding tobacco) or positive urine toxicology.
* Pregnancy (urine pregnancy tests on the day of scans for menstruating girls).
* Inability to provide written informed consent according to the Yale Human Investigation Committee (HIC) guidelines in English.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09-28 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD MS, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Hospital Research Unit at the Yale New Haven Hospital, New Haven, Connecticut
  - Yale Child Study Center, New Haven, Connecticut

REFERENCES:
- [Background] Krystal JH, Karper LP, Seibyl JP, Freeman GK, Delaney R, Bremner JD, Heninger GR, Bowers MB Jr, Charney DS. Subanesthetic effects of the noncompetitive NMDA antagonist, ketamine, in humans. Psychotomimetic, perceptual, cognitive, and neuroendocrine responses. Arch Gen Psychiatry. 1994 Mar;51(3):199-214. doi: 10.1001/archpsyc.1994.03950030035004. PMID 8122957
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Niciu MJ, Ionescu DF, Richards EM, Zarate CA Jr. Glutamate and its receptors in the pathophysiology and treatment of major depressive disorder. J Neural Transm (Vienna). 2014 Aug;121(8):907-24. doi: 10.1007/s00702-013-1130-x. Epub 2013 Dec 8. PMID 24318540
- [Background] Ballard ED, Ionescu DF, Vande Voort JL, Niciu MJ, Richards EM, Luckenbaugh DA, Brutsche NE, Ameli R, Furey ML, Zarate CA Jr. Improvement in suicidal ideation after ketamine infusion: relationship to reductions in depression and anxiety. J Psychiatr Res. 2014 Nov;58:161-6. doi: 10.1016/j.jpsychires.2014.07.027. Epub 2014 Aug 12. PMID 25169854
- [Derived] Lineham A, Avila-Quintero VJ, Bloch MH, Dwyer J. Exploring Predictors of Ketamine Response in Adolescent Treatment-Resistant Depression. J Child Adolesc Psychopharmacol. 2024 Mar;34(2):73-79. doi: 10.1089/cap.2023.0047. Epub 2024 Jan 3. PMID 38170185
- [Derived] Lineham A, Avila-Quintero VJ, Bloch MH, Dwyer J. The Relationship Between Acute Dissociative Effects Induced by Ketamine and Treatment Response in Adolescent Patients with Treatment-Resistant Depression. J Child Adolesc Psychopharmacol. 2023 Feb;33(1):20-26. doi: 10.1089/cap.2022.0086. PMID 36799961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents (aged 13 to 17 years old) were recruited via (1) physician referral or (2) via direct inquiries from families via ClinicalTrials.gov listing. Subjects were enrolled at the Yale Child Study Center (New Haven, CT) between May 2016 and September 2018.
Pre-assignment Details: Participants were to remain on stable dosing of their current medication regimen for the four weeks prior to the first infusion, and during the four-week trial itself. All participants underwent a physical examination, laboratory screening, and electrocardiography.
Groups:
- Ketamine First Then Midazolam: Participants received a Ketamine infusion under blinded conditions, followed by a Midazolam infusion 14 days later. The subject were monitored continuously during both infusions, and every hour for three hours after the infusion and then followed clinically for two weeks.
  Ketamine was infused at a dose of 0.5mg/kg over 40 minutes and midazolam was infused at a dose of 0.045mg/kg over 40 minutes on the Hospital Research Unit of YNHH.
- Midazolam First Then Ketamine: Participants received a midazolam infusion under blinded conditions, followed by a ketamine infusion 14 days later. The subject were monitored continuously during both infusions, and every hour for three hours after the infusion and then followed clinically for two weeks.
  Midazolam was infused at a dose of 0.045mg/kg over 40 minutes and ketamine was infused at a dose of 0.5mg/kg over 40 minutes on the Hospital Research Unit of YNHH.
Period: Overall Study
Arm/Group | Ketamine First Then Midazolam | Midazolam First Then Ketamine
Started | 6 | 11
Completed | 5 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Received Ketamine in the First Infusion: Participants that were randomly assigned to receive a dose of 0.5 mg/kg of Ketamine to be administered Intravenously during 40 minutes in the Hospital Research Unit of YNHH. Participants were monitored continuously during the procedure, and every hour for three hours after the infusion.
- Received Midazolam in the First Infusion: Participants that were assigned to receive a dose of 0.045mg/kg of Midazolam, administered Intravenously during 40 minutes in the Hospital Research Unit of YNHH. Participants were monitored continuously during the procedure, and every hour for three hours after the infusion
- Total: Total of all reporting groups
Arm/Group | Received Ketamine in the First Infusion | Received Midazolam in the First Infusion | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 11 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15.3 [13 to 17] | 15.6 [13 to 17] | 15.4 [13 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 9 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Score for the Montgomery-Asberg Depression Rating Scale sc ore [Mean (Standard Deviation); unit: units on a scale] — Higher scores in this scale indicate more severe depression; each item yields a score of 0 to 6. Clinical judgment determines the rate on the defined scale steps 0, 2, 4, 6 points or between them1, 3, 5 points, denoted as Worsening symptoms.
  It questions the following symptoms:Apparent sadness, Reported sadness, Inner tension, Reduced sleep, Reduced appetite, Concentration difficulties, Lassitude, Inability to feel, Pessimistic thoughts, Suicidal thoughts.
  Usual cutoff are:0 to 6 normal /symptom absent;7 to 19 mild depression; 20 to 34 moderate depression and >34 severe depression.
  units on a scale | 35.6 (7.1) | 31.8 (10.2) | 32.9 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale Score 1 Day After Infusion
Description: Depressive symptoms (measured by Montgomery-Asberg Depression Rating Scale, revised (MADRS) score) on 1 day after infusion, for the cohort of subjects enrolled in the MDD arm of this trial.
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  Usual cutoff points are:
  0 to 6 - normal /symptom absent. 7 to 19 - mild depression. 20 to 34 - moderate depression. >34 - severe depression.
Time Frame: 1 day after the infusion
Population: A total of 17 patients were randomized to receive either Ketamine or Midazolam in the first infusion, one participant in withdrew from the trail after the first infusion because of improvement in her depressive symptoms and did not receive the second infusion.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Ketamine: Participants were randomly be assigned to receive a dose of 0.5 mg/kg of Ketamine (administered intravenously over 40 minutes with a maximum total dose allowed in this study will be 50mg). The participants were monitored continuously during the procedure, and every hour for three hours after the infusion.
  Followed up clinically for the next 2 weeks.
- Midazolam: Participants were assigned to receive a dose of 0.045mg/kg of Midazolam (administered Intravenously over 40 minutes with a the maximum total dose allowed in this study of 4.5mg), The participants were monitored continuously during the procedure, and every hour for three hours after the infusion.They were followed clinically for two weeks.
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 16 | 16
units on a scale | 15.44 [10.51 to 20.37] | 24.13 [18.21 to 30.04]

ADVERSE EVENTS:
Time Frame: 1 hour after after infusion.
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 15/17 | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=17) | Midazolam (N=16)
Feeling like I am in a dream (Nervous system disorders) | 15 (15) | 1 (1)
Spaced out (Nervous system disorders) | 14 (14) | 13 (13)
Disconnected from body (Nervous system disorders) | 12 (12) | 2 (2)
Feeling like thigs are in slow motion (Nervous system disorders) | 11 (11) | 1 (1)
Body parts feel large or small (Nervous system disorders) | 11 (11) | 0 (0)
Time is moving quickly (Nervous system disorders) | 11 (11) | 1 (1)
Feeling like you are in a movie or are a robot (Nervous system disorders) | 9 (9) | 1 (1)
Objects appear different (Nervous system disorders) | 9 (9) | 0 (0)
Sounds changed (Nervous system disorders) | 9 (9) | 0 (0)
World appears in a fog (Nervous system disorders) | 7 (7) | 1 (1)
Gaps in memory (Nervous system disorders) | 7 (7) | 3 (3)

LIMITATIONS AND CAVEATS:
The small sample size and the smaller number of subjects who were randomized to receive ketamine prior to midazolam.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT02579928/Prot_SAP_000.pdf